CLINICAL TRIAL: NCT00910182
Title: Outcome After Conservative and Surgical Treatment of Splenic Injuries After Blunt Abdominal Trauma. Retrospective Study 2002-2008.
Brief Title: Outcome After Conservative and Surgical Treatment of Splenic Injuries After Blunt Abdominal Trauma.
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Pietro Renzulli MD, Bern University Hospital, Departement of Visceral and Transplant Surgery
Other Study IDs: KEK 07-05-09
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2009-05-29 (Estimated); Status verified 2009-05

CONDITIONS: Splenic Rupture; Abdominal Injuries
Keywords: Splenic rupture; abdominal injuries; Surgery; Angiography; Embolisation; Computed tomography; Classification
MeSH Terms: conditions — Splenic Rupture; Abdominal Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: all adult patients with splenic rupture after blunt abdominal injuries admitted to Bern University Hospital between January 2002 and December 2008 and treated non-operatively
- 2: all adult patients with splenic rupture after blunt abdominal injuries admitted to Bern University Hospital between January 2002 and December 2008 who underwent emergency surgical treatment
  Interventions: Procedure: splenorrhaphy
- 3: all adult patients with splenic rupture after blunt abdominal injuries admitted to Bern University Hospital between January 2002 and December 2008 treated non-operatively plus transcatheter arterial embolisation

INTERVENTIONS:
Procedure: splenorrhaphy — surgical treatment of splenic injuries after blunt abdominal trauma.
  Groups: 2

SUMMARY:
Retrospective study in order to investigate the outcome after conservative (with or without transcatheter arterial embolization) and surgical treatment of splenic injuries.

DETAILED DESCRIPTION:
Background

Splenic injuries after blunt abdominal trauma are treated with increasing frequency without operation. Patients undergo observation and bed rest. In certain circumstances an additional transcatheter arterial embolization is performed. It is uncertain which splenic ruptures (injury grades according to Moore) are best treated non-operatively and which are best treated with an emergency operation. Furthermore the value of organ-preserving surgery (splenorrhaphy) is uncertain. In addition, the importance of transcatheter arterial embolisation is unknown.

Objective

Evaluation of outcome (splenic salvage rate, complications, survival) after conservative and surgical treatment. Evaluation of the importance of organ-preserving surgery and of transcatheter arterial embolization.

Methods

All adult patients with splenic injuries after blunt abdominal trauma are included (2002-2008). The patients charts are studied and the following main information retrieved: age, gender, mechanism of accident, grade of splenic injury, concomitant injuries, patient management in the emergency department (fluid administration etc.), diagnostic methods (ultrasound, computed tomography), treatment modalities (bed rest, surgery, embolization), complications of treatment, re-operations, long-term outcome.

ELIGIBILITY:
Inclusion Criteria:

* traumatic splenic rupture
* 16 years and older

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients suffering from traumatic splenic rupture admitted to Bern University Hospital between January 2002 and December 2008
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2002-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Splenic salvage rate | Routine follow-up examinations were performed 3 and 6 months after splenic injury. All patients and/or their treating physicians will be contacted in order gather information about the present health status

SECONDARY OUTCOMES:
Rate of organ-preserving surgery | Routine follow-up examinations were performed 3 and 6 months after splenic injury. All patients and/or their treating physicians will be contacted in order gather information about the present health status
Percentage of secondary splenic ruptures | Routine follow-up examinations were performed 3 and 6 months after splenic injury. All patients and/or their treating physicians will be contacted in order gather information about the present health status
Percentage of patients undergoing a non-operative management | Routine follow-up examinations were performed 3 and 6 months after splenic injury. All patients and/or their treating physicians will be contacted in order gather information about the present health status
Percentage of patients undergoing transcatheter arterial embolisation | Routine follow-up examinations were performed 3 and 6 months after splenic injury. All patients and/or their treating physicians will be contacted in order gather information about the present health status

CONTACTS AND LOCATIONS:
Overall Officials: Pietro Renzulli, MD, Principal Investigator — Bern University Hospital, 3010 Bern, Switzerland
Locations (1):
- Dep. of visceral and transplant surgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Pachter HL, Spencer FC, Hofstetter SR, Liang HG, Hoballah J, Coppa GF. Experience with selective operative and nonoperative treatment of splenic injuries in 193 patients. Ann Surg. 1990 May;211(5):583-9; discussion 589-91. doi: 10.1097/00000658-199005000-00008. PMID 2339919
- [Background] Pachter HL, Guth AA, Hofstetter SR, Spencer FC. Changing patterns in the management of splenic trauma: the impact of nonoperative management. Ann Surg. 1998 May;227(5):708-17; discussion 717-9. doi: 10.1097/00000658-199805000-00011. PMID 9605662
- [Background] Watson GA, Rosengart MR, Zenati MS, Tsung A, Forsythe RM, Peitzman AB, Harbrecht BG. Nonoperative management of severe blunt splenic injury: are we getting better? J Trauma. 2006 Nov;61(5):1113-8; discussion 1118-9. doi: 10.1097/01.ta.0000241363.97619.d6. PMID 17099516
- [Background] Peitzman AB, Heil B, Rivera L, Federle MB, Harbrecht BG, Clancy KD, Croce M, Enderson BL, Morris JA, Shatz D, Meredith JW, Ochoa JB, Fakhry SM, Cushman JG, Minei JP, McCarthy M, Luchette FA, Townsend R, Tinkoff G, Block EF, Ross S, Frykberg ER, Bell RM, Davis F 3rd, Weireter L, Shapiro MB. Blunt splenic injury in adults: Multi-institutional Study of the Eastern Association for the Surgery of Trauma. J Trauma. 2000 Aug;49(2):177-87; discussion 187-9. doi: 10.1097/00005373-200008000-00002. PMID 10963527
- [Background] Harbrecht BG, Peitzman AB, Rivera L, Heil B, Croce M, Morris JA Jr, Enderson BL, Kurek S, Pasquale M, Frykberg ER, Minei JP, Meredith JW, Young J, Kealey GP, Ross S, Luchette FA, McCarthy M, Davis F 3rd, Shatz D, Tinkoff G, Block EF, Cone JB, Jones LM, Chalifoux T, Federle MB, Clancy KD, Ochoa JB, Fakhry SM, Townsend R, Bell RM, Weireter L, Shapiro MB, Rogers F, Dunham CM, McAuley CE. Contribution of age and gender to outcome of blunt splenic injury in adults: multicenter study of the eastern association for the surgery of trauma. J Trauma. 2001 Nov;51(5):887-95. doi: 10.1097/00005373-200111000-00010. PMID 11706335